CLINICAL TRIAL: NCT04872660
Title: Efficacy and Safety of Gushen Antai Pill on Ongoing Pregnancy Rate in Women With Normal Ovarian Reserve Undergoing in Vitro Fertilization Embryo Transfer: A Prospective, Multicentre, Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Efficacy and Safety of Gushen Antai Pill on Ongoing Pregnancy Rate in Women With Normal Ovarian Reserve Undergoing IVF-ET
Acronym: GSATP-FreET
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jing-Yan Song, Principal Investigator, Shandong University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SDUTCMSZG770214
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Female
Keywords: Traditional Chinese Medicine; In vitro fertilization-embryo transfer; Gushen Antai Pill; Normal ovarian reserve; Ongoing pregnancy rate
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GSATP group (Experimental): Gushen Antai Pill (GSATP, 6g* 9 bags, Beijing boran Pharmaceutical Inc.) was required to be taken orally, 6g three times daily combined with vaginal progesterone (90 mg/day Crinone, Merck) from the day of embryo transfer until 10th gestational week.
  Interventions: Drug: Gushen Antai Pill
- Placebo group (Placebo Comparator): Placebo pill is made up of a certain amount of starch and glucose, and is shaped like GSATP according to the National Drug Standards of the State Food and Drug Administration of China. Placebo pill was required to be taken orally, 6g three times daily combined with vaginal progesterone (90 mg/day Crinone, Merck) from the day of embryo transfer until 10th gestational week.
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Gushen Antai Pill — The Gushen Antai Pill (GSATP, Z20030144) is composed of 10 herbs including radix-polygoni multiflori, radix rehmanniae praeparata, cistanche salsa, radix dipsaci, uncaria, semen cuscutae, rhizoma atractylodis macrocephalae, radix scutellariae, radix paeoniae lactiflorae. Its production follows GMP standards and takes the form of water honey pills, each bag of 6g.
  Arms: GSATP group
Drug: Placebo pill — The placebo pill is produced by Beijing boran Pharmaceutical Co., Ltd. It can simulate the appearance, color and smell of GSATP formula, but it has no clinical effect because it has no active ingredients.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to investigate whether oral Gushen Antai pills supplementation for luteal phase support will improve ongoing pregnancy rate in women with normal ovarian reserve in fresh embryo transfer cycles.

DETAILED DESCRIPTION:
Infertility is a growing reproductive health problem, and it is estimated that approximately 15% of couples of reproductive ages are affected. The invention and popularity of IVF-ET technology, although improving sperm egg encounter and fertilization barriers and implanting early embryos from the uterine cavity in vitro, still do not solve the problem of the uterine implantation environment or endometrial receptivity, and the pregnancy rate needs to be further improved. However, traditional Chinese medicine (TCM) has an original theoretical understanding and exact efficacy for gynecological diseases, therefore, it is necessary to supplement TCM interventions with endometrial receptivity as described above.

TCM is a kind of traditional treatment method with thousands of years history in China, and some previous studies have shown its unique experience in assisting pregnancy and reduce vaginal bleeding in early pregnancy . Similar to the notion of "hypothalamus- pituitary-ovary axis" that is established by Western medicine, TCM also has deeply studied the reproductive regulation of kidney and proposed the concept of "kidney-Tian Gui-Chong Ren-uterine axis." According to TCM, "Kidney Governs Reproduction," and female infertility is closely related to kidney deficiency, and the main therapeutic principle of it involves tonification of the kidney.

GSATP is widely used as an adjunctive therapy in women with threatened abortion in China and the clinical effects reflected by the patients remained satisfactory. The function of GSATP is nourishing yin and tonifying the kidney, strengthening Chong and prevent miscarriage. GSATP is used in the early threatened abortion, which belongs to the kidney yin deficiency syndrome of traditional Chinese medicine. GSATP is made up of Dodder, uncaria, Scutellaria, Atractylodes macrocephala, white peony, rehmannia, Polygonum multiflorum, Dipsacus, Cistanche deserticola, mulberry parasitism. The main components of GSATP include baicalin, Atractylodes macrocephala polysaccharide, flavonoids from Cuscuta chinensis, rhynchophylline, polysaccharides, Cistanche polysaccharides, stilbene glycosides and anthraquinone glycosides and triterpenoid saponins, etc. Modern pharmacological studies have found that these ingredients can improve vascular function, regulate immune activity, inhibit uterine contraction and improve ovarian endocrine function, so GSATP may play a role in promoting embryo implantation and preventing pregnancy. However, to improve the success rate of embryo implantation is a complex process and has not been fully studied. Therefore, in treating complex diseases, multi-targeted therapy such as TCM might have unique advantages over western medicine treatment alone. Although GSATP is associated with very good response in patients, lack of high-quality evidence-based medicine has restricted its promotion. The combination of evidence-based medicine, modern medicine and traditional Chinese medicine is a huge field that involves continuous attention and efforts.

GSATP dramatically increased the ongoing pregnancy rate and decreased the prevalence of vaginal bleeding in patients undergoing frozen thawed embryo transfer in our previous study. Recently, it was demonstrated that luteal support combined with GSATP could dramatically increase embryo implantation and clinical pregnancy rates, as well as early pregnancy loss rates, in IVF-ET fresh embryo transfer cycles. However, the study's methodological deficiencies prevented it from reaching a definitive conclusion about GSATP's treatment effect. This was mostly attributed to the unspecified randomization process, the absence of distribution concealment and blinding, no placebo control, and vague inclusion and exclusion criteria. As a result, a well-designed randomized clinical trial is essential to estimate the efficiency and safety of GSATP in optimizing reproductive outcomes in women with normal ovarian reserve during fresh embryo transfer cycles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal ovarian function reserve (5 ≤ AFC ≤ 15, 1.2 ng/ml ≤ AMH ≤ 3.5 ng/ml).
* Patients with regular menstrual cycle (21-35 days) and normal ovulation.
* Initial IVF / ICSI treatment.
* At least one embryo or blastocyst available for transfer.

Exclusion Criteria:

* Age ≥ 43 years old.
* Body mass index (BMI) ≥ 28 Kg/m2.
* "Freeze-all" strategy.
* Those using the natural cycle or mild stimulation for IVF/ICSI treatment.
* Individuals with severe hyperstimulation ovarian syndrome during controlled ovarian stimulation.
* Acceptors of donated oocytes or performed either In vitro Maturation (IVM) or blastocyst biopsy for Preimplantation Genetic Diagnosis (PGD) or Preimplantation Genetic Testing for Aneuploidies (PGT-A).
* History of two or more previous consecutive spontaneous abortions.
* History of two or more previous IVF-ET failures.
* Karyotype abnormalities.
* Polycystic ovary syndrome.
* Presence of a non-surgically treated hydrosalpinx, uterine cavity fluid or endometrial polyp and an ovarian endometriosis cyst requiring surgery, during ovarian stimulation.
* Congenital or acquired abnormalities of uterine anatomy.
* Combined contraindications to assisted reproductive technology or pregnancy, such as uncontrolled abnormalities of liver and kidney function, diabetes mellitus (glycosylated haemoglobin ≤7%, fasting blood glucose <10 mmol/L ), hypertension, thyroid disease, symptomatic heart disease, moderate to severe anaemia, history of malignancy or thromboembolism or propensity to thrombosis, severe psychiatric disorder, acute infections of the genitourinary system, sexually transmitted diseases, serious adverse habits such as drug abuse, exposure to teratogenic amounts of radiation, toxins, or drugs (such as prednisone or other hormones, adrenaline, antibiotics, or hypertension, cardiovascular, or antiviral medications) during the active procedure period , and uterine factor infertility or physical illness which prevents the ability to bear a pregnancy.

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 10 weeks after the day of embryo transfer
  A fetal heartbeat detected by transvaginal ultrasonography over 12 gestational weeks. [Detected via ultrasound]

SECONDARY OUTCOMES:
Positive pregnancy rate | 2 weeks after the day of embryo transfer
  Serum β-hCG level ≥ 10mIU/mL, 14 days after embryo transfer. [Detected via ELISA]
Embryo implantation rate | 3 weeks after the day of embryo transfer
  The number of intrauterine gestational sacs observed divided by the number of embryos transferred. [Detected via ultrasound]
Clinical pregnancy rate | 4 weeks after the day of embryo transfer
  An intrauterine gestational sac with fetal heartbeat detected by transvaginal ultrasonography. [Detected via ultrasound]
Ectopic pregnancy rate | 4 weeks after the day of embryo transfer
  A pregnancy in which implantation takes place outside the uterine cavity. [Detected via ultrasound]
Pregnancy loss rate | 10 weeks after the day of embryo transfer
  Clinically recognized spontaneous loss of pregnancy before the completion of twelve gestational weeks. [Detected via ultrasound]
Multiple pregnancy rate | 10 weeks after the day of embryo transfer
  There were two or more simultaneous fetuses in the uterine cavity. [Detected via ultrasound]
The prevalence of pregnancy constipation | 10 weeks after the day of embryo transfer
  Functional constipation as the presence of at least two out of six symptoms: straining, lumpy or hard stools, a sensation of incomplete evacuation, a sensation of anorectal obstruction/blockage, manual manoeuvres to facilitate defecation and fewer than three spontaneous bowel movements per week. Symptoms must be present at 25% of the defecations and last at least one months. [Evaluated via questionnaire]
The prevalence of threatened abortion | 10 weeks after the day of embryo transfer
  Abdominal pain and vaginal bleeding happened in the first trimester, but the intrauterine fetus still survived. [Detected via ultrasound]
Live birth rate | Beyond 24 weeks of gestation
  Live birth, defined as the birth of at least one child with breath and heartbeat.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inhorn MC, Patrizio P. Infertility around the globe: new thinking on gender, reproductive technologies and global movements in the 21st century. Hum Reprod Update. 2015 Jul-Aug;21(4):411-26. doi: 10.1093/humupd/dmv016. Epub 2015 Mar 22. PMID 25801630
- [Background] Ried K. Chinese herbal medicine for female infertility: an updated meta-analysis. Complement Ther Med. 2015 Feb;23(1):116-28. doi: 10.1016/j.ctim.2014.12.004. Epub 2015 Jan 3. PMID 25637159
- [Background] Smith CA, Armour M, Ee C. Complementary Therapies and Medicines and Reproductive Medicine. Semin Reprod Med. 2016 Mar;34(2):67-73. doi: 10.1055/s-0035-1571194. Epub 2016 Feb 11. PMID 26866600
- [Background] Shen L-H. Observation on the effect of Gushen Antai pill combined withprogesterone on Early Threatened Abortion [in Chinese]. Chin J Maternal Child HealthCare. 2012; 27:4628-9
- [Background] Qin D-N, She B-R, She Y-C. Effects of Flavonoids from Cuscuta chinensis on reproductivefunction of experimental animals and human villi [in Chinese]. Chin J New Drugs Clin Pharmacol. 2000; 11(6):349-51.
- [Background] Chen W-X, Chen S-H, Li W-J, Shu Q, Jiang D-Q. Modern pharmacological study on the sedative effect of baicalein andAtractylodes macrocephala [in Chinese]. J Clin Rational Drug Use. 2012; 5(12B):177-8.
- [Background] Ma B. Research progress on hypotensive effect and mechanism of Uncariarhynchophylla [in Chinese]. China Med Guide. 2011; 8(7):12-4.
- [Background] Wang P. Modern pharmacological research and clinical application of Rehmannia glutinosa [in Chinese]. Modern Distance Educ Trad Chin Med China. 2008; 6(8):986
- [Background] Cao XL, Song JY, Zhang XX, Chen YH, Teng YL, Liu HP, Deng TY, Sun ZG. Effects of a Chinese Patent Medicine Gushen'antai Pills on Ongoing Pregnancy Rate of Hormone Therapy FET Cycles: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Front Endocrinol (Lausanne). 2020 Sep 23;11:581719. doi: 10.3389/fendo.2020.581719. eCollection 2020. PMID 33071986
- [Background] Lu Y, Long XL. Clinical efficacy of Gushen Antai pill combined with progesterone after in vitro fertilization and embryo transfer [in Chinese]. Maternal and Child Health Care of China. 2017;32(9):1980-2.
- [Derived] Xu Y, Hu X, Ai KL, Sun ZG, Song JY. Integrating Chinese Herbal Medicine in IVF: A Protocol for Randomized Controlled Trial of Gushen Antai Pill. Int J Womens Health. 2025 Nov 25;17:4855-4866. doi: 10.2147/IJWH.S554939. eCollection 2025. PMID 41322369
- [Derived] Xu Y, Hu X, Ai KL, Sun ZG, Song JY. Gushen Antai pill for expected normal ovarian responders undergoing IVF-ET (GSATP-FreET): interim analysis of a randomized controlled trial. Contracept Reprod Med. 2025 Mar 13;10(1):19. doi: 10.1186/s40834-025-00352-9. PMID 40082945